CLINICAL TRIAL: NCT02871544
Title: Predictive Value of Dynamic Combination of B-type Natriuretic Peptide and Neutrophil Gelatinase-associated Lipocalin for the Prognosis of Patients With Sepsis
Brief Title: Predictive Value of Dynamic Combination of BNP and NGAL for the Prognosis of Patients With Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Chun Pan, Dr, Zhongda Hospital
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: Zhongda Hospital AKI
Record Dates: First submitted 2016-07-25; First posted 2016-08-18 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: 28-day Mortality; Sepsis
Keywords: BNP; NGAL; Sepsis; Mortality
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low BNP and Low NGAL Group (Sham Comparator): BNP≤100pg/ml and NGAL≤153pg/ml
  Interventions: Other: BNP and NGAL
- High BNP and Low NGAL Group (Active Comparator): BNP>100pg/ml and NGAL≤153pg/ml
  Interventions: Other: BNP and NGAL
- Low BNP and High NGAL Group (Active Comparator): BNP≤100pg/ml and NGAL>153pg/ml
  Interventions: Other: BNP and NGAL
- High BNP and High NGAL Group (Active Comparator): BNP>100pg/ml and NGAL>153pg/ml
  Interventions: Other: BNP and NGAL

INTERVENTIONS:
Other: BNP and NGAL

SUMMARY:
Objective: to clarify the predictive value of brain natriuretic peptide (BNP) in combination with neutrophil gelatinase associated lipocalin (NGAL) for the prognosis of patients with sepsis.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years and <85 years;
* presence of severe sepsis according to Survival Sepsis Campaign 10;
* all patients voluntarily joined this study with informed consents.

Exclusion Criteria:

* participated in other trials within 30 days before the criteria for this trial were met;
* expected to die within 24 hours;
* pregnant;
* advanced malignancy with life expectancy <6 months;
* history of congestive heart failure;
* chronic renal dysfunction (baseline creatinine >176.8μmol/L); and
* relatives were unwilling to agree to the use of full life support.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2015-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
patient-ventilator synchrony for 30mins | 30mins after the patients involved

SECONDARY OUTCOMES:
the numbers of days in the ICU between day 1 and day 28 | the numbers of days in the ICU until day 28
Mechanical ventilation duration between day 1 and day 28 | days of mechanical ventilation between day 1 and day 28
28-day mortality | 28 days after the patients involved

IPD SHARING:
Plan to Share IPD: Undecided